CLINICAL TRIAL: NCT07262112
Title: Efficacy of Resistance Exercise and an Anti-Inflammatory Diet on Pain, Disease Activity, Functional Status, and Quality of Life in Patients With Rheumatoid Arthritis
Acronym: RED-RA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Berra Yamuç Tanrıöğen (Other)
Responsible Party: Sponsor-Investigator, Berra Yamuç Tanrıöğen, Research Assistant, Balikesir University
Organization: Balikesir University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202405; BAUN-MED-RA-2025 (Other: Balıkesir University)
Record Dates: First submitted 2025-11-16; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Anti-inflammatory Diet; Resistance Exercise; Inflammation
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation | interventions — Exercise; Diet

STUDY DESIGN:
Intervention Model Description: Resistance exercise group
  Anti-inflammatory diet group
  diet and resistance exercise group
  Control group
Masking Description: No masking is applied in this study. Both participants and investigators are aware of the assigned interventions, as the study involves exercise and dietary programs that cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- exercise (Experimental): Participants will undergo supervised strengthening exercises using resistance bands in the Physical Medicine and Rehabilitation unit. Sessions will be conducted 3 days per week, each lasting 1 hour, for a total duration of 6 weeks under physician supervision
  Interventions: Behavioral: Exercise
- Diet+exercise (Experimental): Participants will follow a dietitian-supervised anti-inflammatory diet for 3 months. In addition, they will undergo supervised strengthening exercises using resistance bands in the Physical Medicine and Rehabilitation unit. Exercise sessions will be performed 3 days per week, each lasting 1 hour, for a total duration of 6 weeks under physician supervision
  Interventions: Behavioral: Exercise; Behavioral: Diet
- diet (Experimental): Participants will follow a dietitian-supervised anti-inflammatory diet for a duration of 3 months
  Interventions: Behavioral: Diet
- control (Active Comparator): Participants will continue to receive standard medical treatment for rheumatoid arthritis as prescribed by their treating physician. No study-specific intervention will be added, and routine RA medications and management will be maintained throughout the study period
  Interventions: Other: Medical management/current medications per standard of care by personal physician.

INTERVENTIONS:
Behavioral: Exercise — Supervised strengthening exercises using resistance bands in the Physical Medicine and Rehabilitation unit, in addition to participants' standard medical treatment for rheumatoid arthritis. Each session lasts 1 hour and is conducted 3 days per week for a total of 6 weeks under physician supervision. The intervention focuses on improving muscular strength and physical function. Every 3 sessions, the resistance will be increased for participants who do not experience pain after the exercise session.
  Arms: Diet+exercise; exercise
Behavioral: Diet — Dietitian-supervised anti-inflammatory diet followed for 3 months, in addition to participants' standard medical treatment for rheumatoid arthritis. Participants receive individualized dietary counseling and meal plans tailored to reduce inflammation, and adherence to the diet is monitored throughout the study period
  Arms: Diet+exercise; diet
Other: Medical management/current medications per standard of care by personal physician. — Participants continue standard medical treatment for rheumatoid arthritis as prescribed by their physician. No study-specific intervention is added
  Arms: control

SUMMARY:
This study aims to examine how resistance exercises and an anti-inflammatory diet affect pain, daily functioning, disease activity, and quality of life in people with rheumatoid arthritis. Participants will follow a structured exercise program and a diet plan designed to reduce inflammation. The study will measure changes in pain levels, mobility, overall health, and disease symptoms over time. The goal is to determine whether combining exercise and an anti-inflammatory diet can help improve the daily lives and well-being of individuals living with rheumatoid arthritis.

DETAILED DESCRIPTION:
This study examines the combined effects of resistance exercise and an anti-inflammatory diet on clinical outcomes in individuals with rheumatoid arthritis (RA). RA is a chronic inflammatory condition that commonly leads to persistent pain, reduced physical function, and diminished quality of life. Non-pharmacological strategies, including structured exercise and dietary modification, have shown promise as complementary approaches to routine RA management.

Participants in this study will engage in a supervised resistance exercise program along with an anti-inflammatory diet designed to reduce systemic inflammation and support overall musculoskeletal health. The exercise component focuses on improving muscle strength, joint stability, and functional performance, while the dietary intervention emphasizes foods known to lower inflammatory activity.

Outcome assessments will be conducted at baseline (week 0), week 6, and month 3 to evaluate the progression of clinical improvements. Measures will include quality of life, disease activity, functional status, and pain levels. Validated tools and standardized assessment instruments will be used to ensure precise and reliable data collection across all time points.

The aim of this study is to determine whether combining resistance exercise with an anti-inflammatory diet results in meaningful, measurable improvements over time in individuals living with rheumatoid arthritis. The findings may contribute to evidence supporting the integration of multimodal lifestyle interventions into routine RA care.

ELIGIBILITY:
Inclusion Criteria:

* Participant voluntarily agrees to participate in the study and provides written informed consent.
* Aged 18 years or older.
* Has low to moderate disease activity (e.g., according to DAS28 score)

Exclusion Criteria:

* Participants under 18 years of age.
* Uncontrolled diabetes or other metabolic/endocrine disorders.
* Uncontrolled hypertension.
* Any changes in medication within the last 1 month.
* Morbid obesity (BMI > 40).
* Pregnancy.
* Chronic kidney disease.
* Presence of psychiatric disorders.
* Alcoholism.
* Any condition contraindicating exercise, including congestive heart failure, lung disease, cancer, active infection, recent fracture, or recent ligament/tendon injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life | Baseline, 6 weeks, 3 months
  Health-related quality of life will be assessed using Arthritis Impact Measurement Scales 2 (AIMS2) at baseline, 6 weeks, and 3 months. This outcome measure the effect of the study interventions, in addition to participants' standard medical treatment for rheumatoid arthritis A patient-reported questionnaire assessing the physical, emotional, and social impact of arthritis. Scores are calculated for each subscale and overall. Higher scores indicate greater disability or worse health status.
  Units of Measure: points (scale-specific) Minimum Value: 0 points (no impact) Maximum Value: 10 points per subscale (worst impact; total score depends on number of subscales)
change in pain score | Baseline, 6 weeks, 3 months
  Pain will be assessed using the Visual Analog Scale (VAS) at baseline, 6 weeks, and 3 months. This outcome measures the effect of the interventions (Exercise, Diet, Diet+Exercise) in addition to standard medical treatment on patient-reported pain intensity.
  Self-reported measure of pain intensity using a 100-mm horizontal line, where 0 mm represents "no pain" and 100 mm represents "worst imaginable pain." Higher scores indicate greater pain intensity.
  Units of Measure: millimeters (mm) Minimum Value: 0 mm (no pain) Maximum Value: 100 mm (worst imaginable pain)
Change in Disease Activity | Baseline, 6 weeks, 3 months
  Rheumatoid arthritis disease activity will be measured using the Disease Activity Score 28 (DAS28) at baseline, 6 weeks, and 3 months. This outcome evaluates the effect of the interventions combined with standard medical treatment on disease progression and inflammation levels Composite index measuring rheumatoid arthritis disease activity based on the number of tender and swollen joints (28 joints), patient global assessment of health, and either erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP). Higher scores indicate higher disease activity.
  Units of Measure: points Minimum Value: 0 (no disease activity) Maximum Value: ~10 (high disease activity)
Change in Physical Function | Baseline, 6 weeks, 3 months
  Functional status will be assessed using the Health Assessment Questionnaire (HAQ) at baseline, 6 weeks, and 3 months. This outcome measures improvement in patient functionality and ability to perform daily activities under the combined interventions and standard medical treatment A patient-reported questionnaire assessing functional ability in daily activities, including dressing, rising, eating, walking, hygiene, reach, grip, and usual activities. Scores range from 0 to 3, with higher scores indicating greater disability or worse functional status.
  Units of Measure: points Minimum Value: 0 points (no disability) Maximum Value: 3 points (severe disability)
Change in Quality of Life | Baseline, 6 weeks, 3 months
  Health-related quality of life will be assessed using Short Form 36 (SF-36) at baseline, 6 weeks, and 3 months. This outcome measure the effect of the study interventions, in addition to participants' standard medical treatment for rheumatoid arthritis A patient-reported questionnaire assessing overall health-related quality of life across 8 domains, including physical functioning, role limitations, bodily pain, general health, vitality, social functioning, emotional role, and mental health. Each domain is scored from 0 to 100, with higher scores indicating better health status or quality of life.
  Units of Measure: points Minimum Value: 0 points (worst health/quality of life) Maximum Value: 100 points (best health/quality of life)

SECONDARY OUTCOMES:
Change in Physical Function | Baseline, 6 weeks, 3 months
  Functional status will be assessed using validated physical performance tests, including handgrip strength. These assessments will be conducted at baseline, Week 6, and Month 3 to evaluate changes in participants' ability to perform daily activities under the study interventions, in addition to standard medical treatment for rheumatoid arthritis.
  Maximal voluntary grip force measured in kilograms using a hand dynamometer to assess overall muscle strength. Higher values indicate greater muscle strength.
  Units of Measure: kilograms (kg) Minimum Value: 0 kg Maximum Value: ~100 kg (depending on population)
Anthropometric Measurements | Baseline, 6 weeks, 3 months
  Body mass index (BMI) will be measured at baseline, Week 6, and Month 3 to evaluate changes in participants' overall body weight relative to height, in response to the study interventions, alongside standard medical treatment for rheumatoid arthritis.
  BMI calculated as weight in kilograms divided by height in meters squared (kg/m²) to assess overall body weight relative to height. Lower or higher BMI may indicate underweight or overweight status.
  Units of Measure: kg/m² Minimum Value: ~10 kg/m² Maximum Value: ~60 kg/m²
Change in Physical Function | baseline, 6 weeks, 3 months
  Functional status will be assessed using validated physical performance tests, including 30-second sit-to-stand test. These assessments will be conducted at baseline, Week 6, and Month 3 to evaluate changes in participants' ability to perform daily activities under the study interventions, in addition to standard medical treatment for rheumatoid arthritis.
  Number of full stands completed from a seated position in 30 seconds to assess lower body muscle strength and functional performance. Higher values indicate better muscle function.
  Units of Measure: repetitions Minimum Value: 0 repetitions Maximum Value: 60 repetitions
Change in Physical Function | baseline, 6 weeks, 3 months
  Functional status will be evaluated using a validated physical performance measure, the 6-minute walk test (6MWT). Assessments will be performed at baseline, Week 6, and Month 3 to monitor changes in participants' ability to carry out daily activities in response to the study interventions, in addition to standard medical treatment for rheumatoid arthritis.
  Distance walked in meters during 6 minutes to assess functional exercise capacity. Higher values indicate better functional capacity.
  Units of Measure: meters (m) Minimum Value: 0 m Maximum Value: ~1000 m
Anthropometric Measurements | baseline, 6 weeks, 3 months
  Waist circumference will be assessed at baseline, Week 6, and Month 3 to monitor changes in central adiposity associated with the study interventions, in addition to standard medical care for rheumatoid arthritis Measurement of abdominal circumference in centimeters to assess central adiposity. Lower values indicate less abdominal fat.
  Units of Measure: centimeters (cm) Minimum Value: 40 cm (approx.) Maximum Value: 150 cm (approx.)
Anthropometric Measurements | baseline, 6 weeks, 3 months
  Body fat percentage will be measured at baseline, Week 6, and Month 3 to evaluate alterations in participants' total body fat under the study interventions, alongside their standard medical treatment for rheumatoid arthritis.
  Percentage of body mass composed of fat, measured by validated methods such as bioelectrical impedance analysis. Lower values indicate less body fat.
  Units of Measure: percent (%) Minimum Value: 5% Maximum Value: 60%
Anthropometric Measurement | Baseline, 6 weeks, 3 months
  Muscle mass percentage will be assessed at baseline, Week 6, and Month 3 to examine changes in lean body mass resulting from the study interventions, in addition to participants' standard medical care.
  Percentage of body mass composed of skeletal muscle, measured by validated methods such as bioelectrical impedance analysis. Higher values indicate greater muscle mass.
  Units of Measure: percent (%) Minimum Value: 20% Maximum Value: 60%

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Şahin, MD, Principal Investigator — Balikesir University

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT07262112/Prot_SAP_000.pdf